CLINICAL TRIAL: NCT06763874
Title: Pilot Study of Usability and Acceptability for the Optimization of a Functional Electrical Stimulator Controlled by Electromyographic Signal for the Rehabilitation of the Upper Limb in Persons Post-stroke
Brief Title: Usability and Acceptability Study of a Functional Electro-stimulator Controlled by Electromyographic Signal (FitFES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RAISE-FITFES-US
Record Dates: First submitted 2024-12-19; First posted 2025-01-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Healthy Health Care Professionals
Keywords: Stroke; Functional electrical stimulation; Feasibility; Usability; Medical device
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A single-session usability study: ten stroke patients and ten experienced healthcare workers will test the device to evaluate its design and operability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One usability session (Experimental): Subjects will use the device as need-based support to perform motor tasks related to activities of daily living
  Interventions: Device: EMG-based FES device

INTERVENTIONS:
Device: EMG-based FES device — One session of one hour to execute task-oriented exercises with the upper limb while wearing the EMG-based FES device. Submission of questionnaires related to usability, acceptance and satisfaction of the device.

SUMMARY:
Functional recovery of the upper limb after a cerebral stroke is one of the major critical issues in rehabilitation. The advent of innovative technologies can be helpful to rehabilitators and intervene where there is no other solution but a clear therapeutic indication. The use of functional electrostimulators can actively and functionally support movements, helping people affected by stroke to complete a motor gesture taking into account their residual capacities.

DETAILED DESCRIPTION:
FitFES is a wearable and non-invasive device that provides continuous stimulation set according to the residual myoelectric activity of hemiparetic muscles. Its bioinspired functioning has been implemented to restore the neurophysiological feedback from the muscles to the central nervous system while performing voluntary movements.

This study aims to assess the usability, acceptability, and satisfaction of this device by post-stroke subjects and healthcare workers.

Ten post-stroke subjects and ten healthy health care workers will be recruited. Participants will take part in a single session where they are going to execute motor tasks of daily living with the support of the FitFES. At the end of session participants will fill out questionnaires.

Collected results will serve as input for further development of the FitFES device, based on the requests and opinions of participants, to obtain a final version of the device that will be used in a randomized controlled study.

ELIGIBILITY:
Stroke Inclusion Criteria:

* Age equal to or greater than 18 years
* Diagnosis of first ischemic or hemorrhagic unilateral stroke for at least two weeks

Stroke Exclusion Criteria

* Mini Mental State Examination (corrected for age and schooling) < 24
* Clinical evidence of visuospatial disorders, ideomotor apraxia, behavioral disorders, neglect, severe visual and auditory sensory disorders that prevent the use of the device
* Major head trauma
* Cardio-respiratory or internal clinical instability
* Pregnancy
* Severe spasticity (Ashworth scale > 3)
* Skin integrity issues on the surface interfaced with the device
* Implanted electronic devices
* Epilepsy
* Severe peripheral neuropathies

Healthy health care professionals inclusion criteria:

* Age equal to or greater than 18 years

Healthy health care professionals exclusion criteria:

* Pregnancy
* Skin integrity issues on the surface interfaced with the device
* Implanted electronic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | At the end of the single test session (the session is 60 minutes)
  The SUS assesses Usability and Acceptability of a device. The SUS consists of a 10 item questionnaire with five response options for respondents, from strongly agree to strongly disagree.
Unified Theory of Acceptance and Use of Technology (UTAUT) | At the end of the single test session (the session is 60 minutes)
  A questionnaire asking how acceptable and easy to use the technological device is. The theoretical model of UTAUT suggests that the actual use of technology is determined by behavioural intention. The perceived likelihood of adopting the technology is dependent on the direct effect of four key constructs, namely performance expectancy, effort expectancy, social influence, and facilitating conditions. The UTAUT examines the acceptance of technology, determined by the effects of performance expectancy, effort expectancy, social influence and facilitating conditions.

SECONDARY OUTCOMES:
Stroke Rehabilitation Motivation Scale (7-item SRMS) | At the end of the single test session (the session is 60 minutes)
  Motivational impact of the rehabilitation approach used The 7-item SRMS was devised from the 28-item SRMS and inquires upon intrinsic and extrinsic motivation domains for rehabilitation. Scores range from 1 to 7 so the total score can range from 7-35 with higher scores indicating higher motivation.
Rating of Perceived Exertion/Borg 6-20 (RPE) | At the end of the single test session (the session is 60 minutes)
  Perception of the overall and of the upper limb stress. The scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort).
Semi-structured interviews | At the end of the single test session (the session is 60 minutes)
  Open-answer questionnaires related to the use of the FES device, its application in rehabilitation and the subjects perception of device usability
Report of adverse events | At the end of the single test session (the session is 60 minutes)
  Organized reporting of adverse events occurring during the use of the device

OTHER OUTCOMES:
Demographic data and professional background information | At the start of the single test session (the session is 60 minutes)
  Age, gender, scholarity, professional background

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Ferrarin, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi Onlus, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Shared data will comprise only IPD used in results publication. Data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication with no end date
Access Criteria: Request should be addressed to the principal investigator or the corresponding author of the publication.

REFERENCES:
- [Background] Doyle S, Bennett S, Fasoli SE, McKenna KT. Interventions for sensory impairment in the upper limb after stroke. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD006331. doi: 10.1002/14651858.CD006331.pub2. PMID 20556766
- [Background] Hatem SM, Saussez G, Della Faille M, Prist V, Zhang X, Dispa D, Bleyenheuft Y. Rehabilitation of Motor Function after Stroke: A Multiple Systematic Review Focused on Techniques to Stimulate Upper Extremity Recovery. Front Hum Neurosci. 2016 Sep 13;10:442. doi: 10.3389/fnhum.2016.00442. eCollection 2016. PMID 27679565
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed Definitions and a Shared Vision for New Standards in Stroke Recovery Research: The Stroke Recovery and Rehabilitation Roundtable Taskforce. Neurorehabil Neural Repair. 2017 Sep;31(9):793-799. doi: 10.1177/1545968317732668. PMID 28934920
- [Background] Bovonsunthonchai S, Hiengkaew V, Vachalathiti R, Vongsirinavarat M, Tretriluxana J. Effect of speed on the upper and contralateral lower limb coordination during gait in individuals with stroke. Kaohsiung J Med Sci. 2012 Dec;28(12):667-72. doi: 10.1016/j.kjms.2012.04.036. Epub 2012 Jul 28. PMID 23217359
- [Background] Hwang YI, Yoon J. Changes in gait kinematics and muscle activity in stroke patients wearing various arm slings. J Exerc Rehabil. 2017 Apr 30;13(2):194-199. doi: 10.12965/jer.1734898.449. eCollection 2017 Apr. PMID 28503532
- [Background] Perini G, Bertoni R, Thorsen R, Carpinella I, Lencioni T, Ferrarin M, Jonsdottir J. Sequentially applied myoelectrically controlled FES in a task-oriented approach and robotic therapy for the recovery of upper limb in post-stroke patients: A randomized controlled pilot study. Technol Health Care. 2021;29(3):419-429. doi: 10.3233/THC-202371. PMID 33386831
- [Background] Jonsdottir J, Thorsen R, Aprile I, Galeri S, Spannocchi G, Beghi E, Bianchi E, Montesano A, Ferrarin M. Arm rehabilitation in post stroke subjects: A randomized controlled trial on the efficacy of myoelectrically driven FES applied in a task-oriented approach. PLoS One. 2017 Dec 4;12(12):e0188642. doi: 10.1371/journal.pone.0188642. eCollection 2017. PMID 29200424
- [Background] Wafa HA, Wolfe CDA, Emmett E, Roth GA, Johnson CO, Wang Y. Burden of Stroke in Europe: Thirty-Year Projections of Incidence, Prevalence, Deaths, and Disability-Adjusted Life Years. Stroke. 2020 Aug;51(8):2418-2427. doi: 10.1161/STROKEAHA.120.029606. Epub 2020 Jul 10. PMID 32646325
- [Background] Li L, Scott CA, Rothwell PM. Association of Younger vs Older Ages With Changes in Incidence of Stroke and Other Vascular Events, 2002-2018. JAMA. 2022 Aug 9;328(6):563-574. doi: 10.1001/jama.2022.12759. PMID 35943470
- [Background] Dmytriw AA, Dibas M, Phan K, Efendizade A, Ospel J, Schirmer C, Settecase F, Heran MKS, Kuhn AL, Puri AS, Menon BK, Sivakumar S, Mowla A, Vela-Duarte D, Linfante I, Dabus GC, Regenhardt RW, D'Amato S, Rosenthal JA, Zha A, Talukder N, Sheth SA, Hassan AE, Cooke DL, Leung LY, Malek AM, Voetsch B, Sehgal S, Wakhloo AK, Goyal M, Wu H, Cohen J, Ghozy S, Turkel-Parella D, Farooq Z, Vranic JE, Rabinov JD, Stapleton CJ, Minhas R, Velayudhan V, Chaudhry ZA, Xavier A, Bullrich MB, Pandey S, Sposato LA, Johnson SA, Gupta G, Khandelwal P, Ali L, Liebeskind DS, Farooqui M, Ortega-Gutierrez S, Nahab F, Jillella DV, Chen K, Aziz-Sultan MA, Abdalkader M, Kaliaev A, Nguyen TN, Haussen DC, Nogueira RG, Haq IU, Zaidat OO, Sanborn E, Leslie-Mazwi TM, Patel AB, Siegler JE, Tiwari A; North American Neurovascular COVID-19 (NAN-C) Consortium & Society of Vascular and Interventional Neurology (SVIN) Investigators. Acute ischaemic stroke associated with SARS-CoV-2 infection in North America. J Neurol Neurosurg Psychiatry. 2022 Apr;93(4):360-368. doi: 10.1136/jnnp-2021-328354. Epub 2022 Jan 25. PMID 35078916
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936